CLINICAL TRIAL: NCT01540162
Title: Open-labelled, Controlled, Parallel Group Study to Assess the Efficacy and Safety of MUTAFLOR in 3 Weeks Treatment for Immunity Improvement in Preterm Infants With 1 Year Follow-up Period
Brief Title: Experience of Mutaflor Suspension Use in Preterm Infants for Immunity Improvement
Acronym: EMSUP
Status: Completed | Type: Observational
Sponsor: Odessa National Medical University (Other)
Responsible Party: Principal Investigator, Mykola L Aryayev, MD PhD, Professor, MD, PhD, Odessa National Medical University
Other Study IDs: NIS MU 1128 AO
Record Dates: First submitted 2012-02-16; First posted 2012-02-28 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-08

CONDITIONS: Neonatal Infection
Keywords: preterm newborn; neonatology; EcN; Nissle; Mutaflor; prophylaxis; infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group I: Patients of group I are exposed to the probiotic Mutaflor: 1 ml once a day during first week of life, and three times per week during the second and third week of life.
- Group II: Patients of group II remain unexposed to the probiotic Mutaflor.

SUMMARY:
EcN has been registered as a medical drug under the brand name Mutaflor® SUSPENSION in Ukraine in 2010. Indications for its clinical use are acute diarrhea in infants and toddlers including those on tube feeding tube, diarrhea in children, prophylactics of pathological colonization in newborns including premature newborns, and improvement of immunity in newborns (mature and premature).

The aim of this trial was to observe efficacy and safety of Mutaflor® SUSPENSION use for immunity improvement in preterm newborn infants

DETAILED DESCRIPTION:
Study design: open-labeled, controlled, parallel group, non-interventional 3-weeks-study with followed prospective observation during 1 week and 1 year follow-up period.

Patients of group I take the probiotic Mutaflor orally in the dose 1 ml once a day during first week of life and three times per week during the second and third week of life. Patients of the group II don't take specific probiotic for immunity strengthening.

ELIGIBILITY:
Inclusion Criteria:

* age 12-24 hours of life;
* 1st degree of prematurity (functionally mature infant, gestational age 35-36 weeks);
* exclusive breast feeding during study;
* both parents must sign and date an informed consent for infant's participation in the study.

Exclusion Criteria:

* perinatal asphyxia ( Apgar score less than 8);
* significant concomitant disease (congenital birth defects, perinatal encephalopathy, TORCH - infections and other infectious disease of newborn, respiratory distress syndrome ets);
* clinically significant changes in blood analyze results (if needed);
* use of other probiotics or prebiotics during the first 28 days of study participation.

Ages: 12 Hours to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm newborns with gestational age of 35-36 weeks
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mykola L Aryayev, Prof MD PhD, Principal Investigator — Odessa National Medical University
Locations (1):
- Maternity House №5, Odesa, Ukraine

REFERENCES:
- [Derived] Aryayev ML, Senkivska LI, Bredeleva NK, Talashova IV. Prophylaxis of acute respiratory infections via improving the immune system in late preterm newborns with E. coli strain Nissle 1917: a controlled pilot trial. Pilot Feasibility Stud. 2018 Apr 23;4:79. doi: 10.1186/s40814-018-0271-y. eCollection 2018. PMID 29713493

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I | Group II
Started | 30 | 32
Completed | 30 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Categorical [Count of Participants; unit: Participants] — Newborns
  Participants
    <=18 years | 30 | 32 | 62
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 16 | 17 | 33
Region of Enrollment [Number; unit: participants]
  Ukraine | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: The Number (Rate) of Patients With Acute Respiratory Infections
Description: ARI: Acute Rhinitis, Acute Rhinopharyngitis, Acute Bronchitis, Acute Bronchiolitis and Pneumonia
Time Frame: first 28 days of life
Measure: Number; unit: participants
Arm/Group | Group I | Group II
Number analyzed (Participants) | 30 | 32
participants | 3 | 14
Statistical Analysis 1: Comparison: Group I vs Group II; Test type: Superiority or Other; p = 0.05, Chi-squared; Risk Ratio (RR) = 0.23, 95% CI 2-sided [0.05 to 0.73]

2. Secondary Outcome: The Number (Rate) of Patients With Acute Respiratory Infections
Description: ARI: Acute Rhinitis, Acute Rhinopharyngitis, Acute Bronchitis, Acute Bronchiolitis and Pneumonia
Time Frame: first 6 month of life
Measure: Number; unit: participants
Arm/Group | Group I | Group II
Number analyzed (Participants) | 30 | 32
participants | 15 | 23

3. Secondary Outcome: The Number (Rate) of Patients With Acute Respiratory Infections
Description: ARI: Acute Rhinitis, Acute Rhinopharyngitis, Acute Bronchitis, Acute Bronchiolitis and Pneumonia
Time Frame: first 12 month of life
Measure: Number; unit: participants
Arm/Group | Group I | Group II
Number analyzed (Participants) | 30 | 32
participants | 23 | 29

ADVERSE EVENTS:
Arm/Group | Group I | Group II
Serious Adverse Events (participants affected / at risk) | 11/30 | 20/32
Other Adverse Events (participants affected / at risk) | 15/30 | 22/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (N=30) | Group II (N=32)
Acute Respiratory and Gastrointestinal Infections (Infections and infestations) | 11 (12) | 20 (22) — Hospitalisation due to ARIs and GIs
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (N=30) | Group II (N=32)
Acute Respiratory Infections (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 22 (24) — acute rhinitis, acute rhinopharyngitis, acute bronchitis
Gastrointestinal disorders (Gastrointestinal disorders) | 12 (14) | 13 (14) — infant colic, acute enterocolitis, constipation, regurgitation, diarrhoea
dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) — diaper dermatitis, atopic dermatitis
Changed Blood Parameter (Blood and lymphatic system disorders) | 2 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No